CLINICAL TRIAL: NCT02601430
Title: Functional Magnetic Resonance Angiographic Imaging Using Blood Oxygen Level Determination (BOLD) Assessment as a Surrogate of Improved Skeletal Muscle Oxygenation After Endovascular Therapy for the Treatment of Chronic Lower Limb Ischemia
Brief Title: BOLD MRI as a Surrogate of Improved Muscle Oxygenation Following Endovascular Therapy for the Treatment of CLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BB-BOLD-15
Record Dates: First submitted 2015-10-30; First posted 2015-11-10 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BOLD-MRI (Experimental): Blood Oxygen Level Dependent (BOLD)-MRI assessment of limb perfusion before and after standard of care endovascular therapy.
  Interventions: Other: BOLD-MRI

INTERVENTIONS:
Other: BOLD-MRI — A fixed air cuff will be placed on the index limb at the level of the calf and will be inflated to a level which induces the loss of the pedal Doppler signal. Inflation will be maintained for 180 seconds, then will be rapidly deflated and BOLD MR imaging will be initiated.

SUMMARY:
The purpose of this study is to determine if an MRI technique called Blood Oxygen Level Dependent, or BOLD, can be used to evaluate blood flow in the leg before and after treatment with standard endovascular therapy in patients with chronic lower limb ischemia.

DETAILED DESCRIPTION:
This study is a prospective single arm, open label registry to evaluate the feasibility of blood oxygen level dependent (BOLD) magnetic resonance imaging for the assessment of a potentially new functional surrogate of altered lower limb skeletal muscle oxygenation after a successful percutaneous endovascular intervention. Baseline MRI assessment using the BOLD technique will be performed on qualified subjects prior to undergoing a standard of care endovascular therapy. Post-procedure BOLD-MRI assessment will also be performed at 30 days and either 90 or 180 days post-procedure. Post-MR image acquisition processing and analysis will be performed, using pre-determined algorithms, by a core laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 90 years
* Subject has been informed of the nature of the study and agreed to participate and has signed an IRB approved consent form
* Subject understands the duration of the study and its follow-up visit requirements and agrees to comply
* Subject has documented chronic limb ischemia in the target limb with Rutherford Category 2-5 and pulse plethysmography (PPG), pulse volume recording (PVRs), TcPO2, ABIs or toe pressures and symptoms that conform to the diagnosis of life-style limiting claudication or critical limb ischemia

Exclusion Criteria:

* Adult subjects who lack the capacity to consent for themselves
* Women who are pregnant or wish to become pregnant during the course of the study. (Women of child-bearing potential must undergo pregnancy testing at the time of enrollment, and be counseled in appropriate measures to avoid becoming pregnant for the duration of the study)
* Subjects with contraindications to MR imaging procedures (including the administration of gadolinium based contrast agents)
* Subjects suspected to be unable to withstand the reactive hyperemia protocol

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Enhanced oxygen reperfusion of the index foot assessed by BOLD MRI before and after endovascular intervention. | 6 months
  The BOLD MR T2* signal will be analyzed pre-and post-endovascular intervention to determine if it is able to detect a difference in foot oxygen perfusion levels.

CONTACTS AND LOCATIONS:
Overall Officials: Krishna J Rocha-Singh, MD, Principal Investigator — St. John's Hospital
Locations (1):
- St. John's Hospital, Springfield, Illinois, United States